CLINICAL TRIAL: NCT04885426
Title: The Role of Metformin in the Prevention for Colorectal Adenoma Recurrence in Post-polypectomy Patients
Brief Title: Metformin for the Prevention of CRA Recurrence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jing-yuan Fang, MD, Ph. D (Other)
Responsible Party: Sponsor-Investigator, Jing-yuan Fang, MD, Ph. D, Director of Department of Gastroenterology, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KY2019-019
Record Dates: First submitted 2020-11-29; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Colorectal Adenoma; Metformin; Chemoprevention
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participant, investigator, data analyst, endoscopist and pathologist involved in this study are all blinded of which treatment the participants are receiving. The pharmaceutical company provided blinded bottles of study pills with the label 'A' , 'B' or 'C'. Unblinding will be advanced only in case of emergency.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low-dose metformin group (Experimental): low-dose metformin, 250mg/day
  Interventions: Drug: low-dose metformin
- high-dose metformin group (Experimental): high-dose metformin, 500mg/day
  Interventions: Drug: high-dose metformin
- control group (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: low-dose metformin — Metformin Pill 250mg/day
  Arms: low-dose metformin group
Drug: high-dose metformin — Metformin Pill 500mg/day
  Arms: high-dose metformin group
Drug: Placebo — Placebo
  Arms: control group

SUMMARY:
Most of the sporadic colorectal cancer (CRC )develop from colorectal adenoma (CRA), patients with CRA have a high risk of recurrence and development of metachronous CRA or CRC after removal, therefore, the investigators conducted this clinical trial to explore the chemoprevetion effect of metformin for CRA recurrence after removal.

DETAILED DESCRIPTION:
Colorectal adenomas are well-known to be precancerous lesions that develop into colorectal cancers on the basis of the adenoma-carcinoma sequence. The effects of screening for colorectal adenomas and removing precancerous lesions on the prevention of colorectal cancer have been established. Because of the high recurrence rates of colorectal adenomas in patients who have undergone polypectomy, the potential chemopreventive agents that may reduce the risk of colorectal adenoma recurrence need to be investigated.

Metformin is a widely used diabetes medicine. In recent years, anticancer activity of metformin has been explored. The aim of this study is to investigate the effect of metformin on the recurrence of colorectal adenomas by conducting a randomized, placebo-controlled, prospective clinical.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 40-80 years without diabetes;
2. CRAs removed without recurrence before recruitment;
3. Must sign the consent form after being fully informed and understanding the purpose and procedure of this study.

Exclusion Criteria:

1. Familial adenomatous polyposis (FAP) or hereditary non-polyposis colorectal cancer (HNPCC, Lynch syndrome);
2. Regularly taking aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs), cyclo-oxygenase 2 (COX2) inhibitors, calcium or vitamin D;
3. Have a history of gastrointestinal surgery;
4. Have severe heart, liver or kidney disease ;
5. Have cancer history;
6. Women with pregnant, during breast-feeding period, or with expect pregnancy;
7. Diabetes（taking diabetes medicines or HbA1c>6.5%);
8. Inflammatory bowel disease;
9. Mental illness;
10. Intolerant to metformin;
11. Cannot tolerate colonoscopy;
12. Staffs in this clinical trial;
13. Poor bowel preparation for colonoscopy or the examination time is shorter than 6 minutes;
14. Unsuitable for inclusion by the investigator

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
CRA recurrence rate | one year, two years
  Percentage of patients who has recurrence of CRA(colorectal adenoma) during or after chemotherapy with metformin or placebo.

SECONDARY OUTCOMES:
All polypoid lesions incidence rate | one year, two years
  Percentage of patients who has incidence of all polypoid lesions during or after chemotherapy with metformin or placebo.
CRC incidence rate | one year, two years
  Percentage of patients who has incidence of CRC (colorectal cancer) during or after chemotherapy with metformin or placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Yuan Fang, Professor, Study Director — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Division of Gastroenterology and Hepatology, Ren-Ji Hospital, Shanghai Jiao-Tong University School of Medicine, Shanghai Institute of Digestive Disease; Key Laboratory of Gastroenterology & Hepatology, Ministry of Health, Shanghai, Shanghai Municipality, China